CLINICAL TRIAL: NCT03936985
Title: Validation of a Community Pharmacy-Based Prescription Drug Monitoring Program Risk Screening Tool
Acronym: PHARMSCREEN
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: University of Cincinnati (Other); Purdue University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jerry Cochran, Associate Professor, University of Utah
Other Study IDs: CTN-0093; 5UG1DA049444 (NIH)
Record Dates: First submitted 2019-04-30; First posted 2019-05-03 (Actual); Results first posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Opioid Abuse; Prescription Drug Abuse (Not Dependent)
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of the study is to validate a Prescription Drug Monitoring Program-based opioid risk metric to discriminate between low, moderate, and high-risk opioid use disorder. The World Health Organization Alcohol, Smoking, and Substance Involvement Screening Test (WHO ASSIST) will be used as the gold standard instrument that defines patient risk levels. No intervention or hypothesis will be tested.

DETAILED DESCRIPTION:
Fatal overdose deaths involving prescription opioids, heroin, and synthetic opioids has continued to increase across the US-continuing to increase in 35 states from 2013-2017. Given these persistent trends for adverse opioid-related outcomes in populations across the US, it is critical to work to identify those who are at risk, deliver appropriate care that will help prevent progression to more severe opioid-related outcomes, and provide referral and treatment resources to those who suffer from opioid use disorder. Therefore, it is necessary to expand the continuum of care to health care settings that previously may have been underutilized. One underutilized resource for addressing the current opioid epidemic is community pharmacies.The most important clinical tool pharmacists have available to identify possible misuse of opioid medications is prescription drug monitoring programs (PDMP),which capture patient-level prescription dispensing information to inform monitoring, dispensing decisions, and possible intervention.These tools are available in all US states and have the potential to enable pharmacists to identify patients at-risk for opioid-related adverse events, such as addiction and overdose. In light of the continued escalation of the opioid epidemic nationally, combined with the promising opportunities afforded by the further inclusion of community pharmacy settings for engaging patients with opioid-related risk, it is important to evaluate whether current PDMP risk metrics correlate with clinically validated opioid risk tools and if clinically meaningful risk cutoffs exist for PDMP risk metrics.

This study will evaluate the concurrent validity of a PDMP-based opioid risk metric as a clinical measure of high risk opioid use and establish clinically useful risk-level thresholds relative to the widely validated gold standard of the World Health Organization Alcohol, Smoking, and Substance Involvement Screening Test (WHO ASSIST). This study is a one group, cross-sectional, health assessment study. Participants who enroll in the study will complete on-line surveys at a single time point. Approximately 1,523 patients will be recruited from approximately 15 community community pharmacies. Trained pharmacy staff will inform potentially eligible participants, or individuals receiving at least one prescription(s) for potentially eligible participants, of the survey opportunity. Patients recruited will complete validated measures to assess opioid use and risk behaviors, substance use, and physical and mental health. A series of a priori analyses will be conducted to evaluate the validity of the PDMP-based opioid risk metric relative to the widely validated gold standard WHO ASSIST and to identify cutoff thresholds. Correlational, regression, and Cohen's Kappa statistical analyses will also be conducted to evaluate the relationship between the risk metric and the WHO ASSIST.

ELIGIBILITY:
Inclusion Criteria:

1. be dispensed ≥1 opioid medication (including tramadol) by a participating pharmacy;
2. be ≥18 years of age according to pharmacy data and self-report

Exclusion Criteria:

1. solely filling buprenorphine or buprenorphine combination products i.e., patients receiving OUD treatment with no other opioid medication use;
2. currently receiving treatment for cancer;
3. having previously completed the survey;
4. having current involvement with the criminal justice system that has, or could, lead to incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults 18 years or older, prescribed opioid medications from one of 15 participating pharmacies.
Sampling Method: Non-Probability Sample
Enrollment: 1464 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Cincinnati, Cincinnati, Ohio
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Charron E, Brooks JH, Peterson KT, Akinwolere OG, Winhusen T, Cochran G. Mapping prescription drug monitoring program data to self-report measures of non-medical prescription opioid use in community pharmacy settings. Res Social Adm Pharm. 2023 Aug;19(8):1171-1177. doi: 10.1016/j.sapharm.2023.04.121. Epub 2023 Apr 23. PMID 37142474
- [Derived] Charron E, Okifuji A, Bryan MA, Reese S, Brown JL, Ferguson A, Ghitza UE, Winhusen T, Cochran G. Pain Severity and Interference and Substance Use Among Community Pharmacy Patients Prescribed Opioids: A Secondary Analysis of the PHARMSCREEN Study. J Pain. 2022 Aug;23(8):1448-1459. doi: 10.1016/j.jpain.2022.03.238. Epub 2022 Apr 11. PMID 35417791

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Study participants were patients of one of the 19 study pharmacies, completed the survey, and had sufficient data in the prescription drug monitoring program to generate the Narcotic Score (NS)
Period: Overall Study
Arm/Group | All Participants
Started | 1464
Completed | 1464
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 1464
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 911
  Male | 553
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 1447
  Unknown or Not Reported | 0
Prescription Opioids [Count of Participants; unit: Participants] — Prescription Opioids is measured using the WHO ASSIST (The Alcohol, Smoking and Substance Involvement Screening Test).
  Participants
    Low | 772
    Moderate | 623
    High | 33
    Unknown/Not responded | 36

OUTCOME MEASURES:

1. Primary Outcome: Validity of the PDMP Narcotic Score Versus the WHO ASSIST
Description: To assess the validity of the PDMP Narcotic Score, the AUC (Area Under the Curve) was used. AUC ranges in value from 0 to 1. A model whose predictions are 100% wrong has an AUC of 0.0; one whose predictions are 100% correct has an AUC of 1.0. And when AUC is 0.5, it means the model has no means of separating between the different groups. For this study, the closer to 1.0 the more similar the PDMP Narcotic Score is to the WHO ASSIST.
Time Frame: The ASSIST was administered once at Day 1.
Population: Participants who complete the World Health Organization Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST).
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- High to Moderate Risk: High- compared to moderate-risk for prescription opioid use on the ASSIST
- Moderate to Low Risk: Moderate- compared to low-risk for prescription opioid use on the ASSIST
Arm/Group | High to Moderate Risk | Moderate to Low Risk
Number analyzed (Participants) | 33 | 1395
probability | .70 [0.59 to 0.80] | .74 [.71 to .76]

ADVERSE EVENTS:
Time Frame: This was a minimal risk study, and as such no adverse events were collected.
Description: All-cause mortality, serious adverse events, and other (not including serious) adverse events were not monitored.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/85/NCT03936985/Prot_002.pdf
  • Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/85/NCT03936985/SAP_003.pdf
  • Informed Consent Form (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/85/NCT03936985/ICF_000.pdf